CLINICAL TRIAL: NCT03284021
Title: A Pilot Study on 1550 nm Fractional Erbium-glass Laser for Alopecia Treatment
Brief Title: Fraxel Laser for Alopecia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study did not start.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology-Head and Neck Surgery, and Surgery, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00205107
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Alopecia
MeSH Terms: conditions — Alopecia | interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fraxel laser (Other)
  Interventions: Device: Fractional erbium-glass 1550 nm laser

INTERVENTIONS:
Device: Fractional erbium-glass 1550 nm laser — The fractional erbium-glass 1550 nm laser will be applied to the previously 100 cm2 determined area of the scalp with the following parameters: 5-10 mm tip, 5-10 mJ, pulse energy 500-1500 MTZ/cm2 density, one to twopasses, static mode.
  Other Names: Fraxel RE:STORE

SUMMARY:
This is a pilot study to evaluate the effect of the 1550 nm fractional erbium-glass laser in patients with nonscarring alopecias. Participants currently living in the Chicago metropolitan area and meet inclusion/exclusion criteria will be considered for enrollment. Participants will receive 5 sessions of laser, 30 days apart, to the area of alopecia on the scalp. Follow-up is at 150 days.

This study was a pilot study designed to determine feasibility of this procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years old
2. Subjects are in good health as judged by the investigator.
3. Diagnosed by a dermatologist with mild to moderate androgenetic alopecia or alopecia areata.
4. Subject is seeking treatment for alopecia.
5. Subject has never previously used finasteride or minoxidil or has consistently used finasteride or minoxidil for at least 1 year.
6. Subjects who are willing and have the ability to understand and provide informed consent for participation in the study and are able to communicate with the investigator.

Exclusion Criteria:

1. Evidence of another skin condition affecting the treatment area that would interfere with clinical assessments.
2. Subjects who are unwilling to avoid initiating treatment with minoxidil or finasteride for the duration of the study; or in subjects who have been treated with minoxidil or finasteride for at least 1 year, unwilling to avoid changes in the dosing regimen of these medications for the duration of the study.
3. Willing to refrain from washing hair or using hair product 24 hours before and after treatment visits
4. History of recurrent facial or labial herpes simplex infection
5. History of hypertrophic scars or keloids
6. Subjects who have any requirement for the use of local or systemic steroids or other immunosuppressive agent
7. Pregnant or breast feeding
8. Uncooperative patients or patients with neurological disorders who are incapable of following directions or who are predictably unwilling to return for follow-up examinations.
9. Subjects who are unable to understand the protocol or give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-24 (Estimated); Primary Completion 2019-04-24 (Estimated); Study Completion 2019-04-24 (Estimated)

PRIMARY OUTCOMES:
Clinical change of alopecia from baseline to 150 days. | Baseline and 150 Days
  Outcome assessors will measure clinical change using the Jaeschke scale, a 15 point scale that describes how worse or better the condition is.

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No